CLINICAL TRIAL: NCT01902082
Title: Phase I Study of Allogeneic Adipose-derived Mesenchymal Stem Cells in Acute Respiratory Distress Syndrome
Brief Title: Adipose-derived Mesenchymal Stem Cells in Acute Respiratory Distress Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaoxing Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MSCs in ARDS
Record Dates: First submitted 2013-07-14; First posted 2013-07-18 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: ARDS
Keywords: ARDS; mesenchymal stem cells; Safety; Cytokines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesenchymal stem cell arm (Experimental): Patients received one dose of 1x 10^6 allogeneic adipose-derived mesenchymal stem cells/kg body weight intravenously within 48 hours of enrollment.
  Interventions: Drug: Mesenchymal stem cells
- Placebo (Placebo Comparator): Patients received one dose of normal saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mesenchymal stem cells
  Arms: Mesenchymal stem cell arm
Drug: Placebo
  Other Names: Intravenous saline infusion will be designated as placebo.
  Arms: Placebo

SUMMARY:
Currently, there is no proven effective pharmacologic treatment available for patients with the acute respiratory distress syndrome (ARDS). Mesenchymal stem cells have been shown to be effective in treating several inflammatory diseases. The main purpose of this study is to assess the safety of allogeneic adipose-derived mesenchymal stem cells in patients with ARDS.

ELIGIBILITY:
Inclusion Criteria:

1. ARDS diagnosed using Berlin definition
2. Eligible patients were at least 18 years of age had acute onset of ARDS.
3. Bilateral opacities in chest radiography
4. No cardiac failure
5. PaO2/FiO2 ratio < 200

Exclusion Criteria:

1. 72 hours after all inclusion criteria met
2. Pre-existing severe diseases of any major organs
3. Pregnancy
4. Pulmonary hypertension
5. Malignant diseases
6. HIV infections.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Compare the adverse events between mesenchymal stem cell treatment and placebo groups | From day 0 at the start of treatment to day 28.

SECONDARY OUTCOMES:
Hospital indices by treatment group | From admission to discharge
  Days in hospital ICU free days at day 28 Ventilator free days at day 28

OTHER OUTCOMES:
cytokines | Day 0 to day 7
  IL-6, IL-8, SP-D, TNF-alpha

CONTACTS AND LOCATIONS:
Locations (1):
- Shaoxing Second Hospital, Shaoxing, Zhejiang, China

REFERENCES:
- [Derived] Zheng G, Huang L, Tong H, Shu Q, Hu Y, Ge M, Deng K, Zhang L, Zou B, Cheng B, Xu J. Treatment of acute respiratory distress syndrome with allogeneic adipose-derived mesenchymal stem cells: a randomized, placebo-controlled pilot study. Respir Res. 2014 Apr 4;15(1):39. doi: 10.1186/1465-9921-15-39. PMID 24708472